CLINICAL TRIAL: NCT06394531
Title: Jaboticaba (Plinia Cauliflora) as a Strategy to Modulate Inflammation, Oxidative Stress, and Gut Dysbiosis in Patients With Chronic Kidney Disease
Brief Title: Effects of Jaboticaba (Plinia Cauliflora) Supplementation in Chronic Kidney Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: DeniseMafra20
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney diseases; jaboticaba; inflammation; oxidative stress; microbitoa
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Jaboticaba peel extract. Patients will ingest 4 capsules/day of jaboticaba (Plinia Cauliflora) peel extract, providing 3.3g of jabuticaba peel extract daily, containing 600mg of phenolic compounds, for one month.
  Interventions: Dietary Supplement: Jaboticaba Peel Extract
- Placebo (Placebo Comparator): Placebo. Patients will ingest 4 capsules/day of placebo (corn starch), providing 3.3g of placebo, for one month.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Jaboticaba Peel Extract — Jaboticaba peel extract. Patients will ingest 4 capsules/day of jaboticaba (Plinia Cauliflora) peel extract, providing 3.3g of jabuticaba peel extract daily, containing 600mg of phenolic compounds, for one month.
  Arms: Intervention
Other: Placebo — Placebo. Patients will ingest 4 capsules/day of placebo (corn starch), providing 3.3g of placebo, for one month.
  Arms: Placebo

SUMMARY:
The increase prevalence of chronic kidney disease (CKD) over the years represent a significant public health problem. The role of inflammation and oxidative stress in the pathophysiology of CKD, as well as progression and comorbidities, is already well consolidated. The gut microbiota composition imbalance may also be a risk factor contributing to the increased conditions mentioned above, and to uremic toxins release and endotoxemia. The literature has indicated the use of bioactive compounds as a nonpharmacological treatment strategies for the management of non-communicable diseases (NCDs), such as CKD and its complications. In this context, jaboticaba (Plinia Cauliflora) emerges as a potential therapeutic approach as it is a source of phenolic compounds, such as anthocyanins, flavonols, ellagitannins, and phenolic acids. Such phenolic compounds may have beneficial effects in patients with CKD, such as anti-inflammatory, antioxidant, modulation of the intestinal microbiota, hypotensive and hypoglycemic effects. These combined effects can help manage risk factors and CKD itself, and associated complications. Therefore, this research project aims to add scientific knowledge, providing a non-pharmacological therapeutic approach to be implemented in clinical practice and in the care of patients with CKD, with the aim of modulating inflammation, oxidative stress, microbiota composition, and improving the quality of life of these patients. Therefore, this study aims to evaluate the effects of jaboticaba (Plinia Cauliflora) supplementation on complications associated with CKD.

DETAILED DESCRIPTION:
This is a chronic study, which consists of a longitudinal, randomized, double-blind, crossover clinical study, with a washout period and placebo-controlled trial. Thirty patients with CKD undergoing hemodialysis will be selected (according to sample calculation, considering p=0.05 and test power of 80%). Randomization will be computerized in a 1:1 ratio, with a block size of 15 (Jaboticaba and Control groups), to receive jaboticaba peel extract or placebo. Eligible patients of both genders, previously evaluated and authorized by the medical and nutritionist team, will be invited to participate in the research in person and verbally, during nutritional consultations at the Prodoctor Hemodialysis Clinic. The intervention consists of supplementing 4 capsules/day, providing 3.3g of jabuticaba peel extract daily, containing 600mg of phenolic compounds, or the same amount of placebo, corn starch, for one month. After the end of this first intervention, blood and fecal samples will be collected again. Followed by a 2-month washout period. After 2 months, blood and fecal samples will be collected again from these patients. The crossover will then begin, the second moment of supplementation in which the patients who received the jaboticaba peel extract in the first moment start to receive the placebo, and the patients who received the placebo initially began to receive jabuticaba peel extract supplementation for one month. At the end of the second supplementation period, blood and fecal samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years
* Clinical diagnosis of Chronic Kidney Disease
* Conservative treatment group: CKD stages 3 and 5 receiving nutritional treatment for at least 6 months
* Hemodialysis group: Hemodialysis patients for more than 6 months

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Autoimmune diseases
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 4 weeks
  Antioxidant and anti-inflammatory biomarker
  Get blood samples to evaluate the supplementation effects in antioxidant and anti-inflammatory biomarker- nuclear receptor factor 2 (Nrf2)
Inflammatory biomarker | 4 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarker- factor nuclear kappa B (NFkB)
Microbiota Composition | 4 weeks
  Get fecal samples to evaluate the supplementation effects in microbiota composition.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, Phd, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lima MDC, do Nascimento HMA, da Silva JYP, de Brito Alves JL, de Souza EL. Evidence for the Beneficial Effects of Brazilian Native Fruits and Their By-Products on Human Intestinal Microbiota and Repercussions on Non-Communicable Chronic Diseases-A Review. Foods. 2023 Sep 19;12(18):3491. doi: 10.3390/foods12183491. PMID 37761200